CLINICAL TRIAL: NCT04972097
Title: Pivotal Study of the NanoKnife System for the Ablation of Prostate Tissue in an Intermediate-Risk Patient Population
Brief Title: Pivotal Study of the NanoKnife System for the Ablation of Prostate Tissue
Acronym: PRESERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ONC-01
Record Dates: First submitted 2021-07-02; First posted 2021-07-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate Tissue; NanoKnife System; Focal Therapy; Intermediate-Risk; Irreversible Electroporation (IRE)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- IRE Treatment Arm (Experimental): All patients enrolled in this trial will receive IRE treatment with the NanoKnife System
  Interventions: Device: Irreversible Electroporation

INTERVENTIONS:
Device: Irreversible Electroporation — IRE of the prostate is typically performed with the subject in the lithotomy position, with 2-6 monopolar probes placed through the perineum using a brachytherapy grid and ultrasound or CT guidance. IRE supplies the targeted tissue with high voltage (2-3 kV) direct current pulses lasting up to 100 microseconds through the electrode probes.
  Other Names: The NanoKnife System

SUMMARY:
Pivotal study to evaluate the use of the NanoKnife System as a focal therapy option for prostate cancer patients. This study will assess the safety and effectiveness of the device when used to ablate prostate tissue in intermediate-risk prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Is greater than 50 years of age
2. Has at least a 10-year life expectancy
3. Has histologically confirmed organ-confined prostate cancer, clinical stage ≤ T2c
4. Has a PSA ≤ 15 ng/mL or PSA density < 0.2 ng/mL2 if PSA is > 15 ng/mL
5. Has Gleason score 3+4 or 4+3
6. Has no evidence of extraprostatic extension by mpMRI
7. Has no evidence of seminal vesicle invasion by mpMRI, and if suspected, confirmed by biopsy
8. Physician is able to visualize prostate gland adequately on transrectal ultrasound imaging during enrollment evaluation
9. Transperineal or transrectal targeted prostate biopsies of lesion, plus 10 core systematic biopsies to include adequate sampling of the peripheral zone correlating with an intermediate risk lesion in the area of the MR-visible lesion
10. A visible lesion on mpMRI that is accessible to Irreversible Electroporation (IRE) treatment (Note: A non-MRI visible lesion detected via systematic standard biopsy will not be considered an exclusion criterion provided the non-MRI visible lesion is singularly located in the contralateral hemisphere of the prostate; is Gleason 6; and comprises no more than 6 mm linear extent of prostate-bearing tissue in a single core on standard biopsy)
11. Has signed a written informed consent and in the judgment of the physician, the study is in the best interest of the subject
12. Understands and accepts the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria:

1. Has known hypersensitivity to pancuronium bromide, atricurium or cisatricurium
2. Is unfit for anesthesia or has a contraindication for agents listed for paralysis
3. Has an active urinary tract infection (UTI)
4. Has a history of bladder neck contracture
5. Is interested in future fertility
6. Has a history (within 3 years) of inflammatory bowel disease
7. Has a concurrent major debilitating illness
8. Had active treatment for a malignancy within 3 years, including malignant melanoma, except for prostate cancer or other types of skin cancer
9. Has any active implanted electronic device (e.g., pacemaker)
10. Is unable to catheterize due to a urethral stricture disease
11. Has had prior or current prostate cancer therapies:

    1. Biologic therapy for prostate cancer
    2. Chemotherapy for prostate cancer
    3. Hormonal therapy for prostate cancer within three months of procedure
    4. Radiotherapy for prostate cancer
    5. Surgery for prostate cancer
12. Has had prior transurethral prostatectomy (TURP), stricture surgery, urethral stent or prostatic implants
13. Has had prior major rectal surgery (except hemorrhoids)
14. Is unfit for pelvic MRI scanning (e.g., severe claustrophobia, permanent cardiac pacemaker, metallic implants that are likely to contribute significant image artifacts, allergy or contraindication to gadolinium (to enhance MRI))
15. Is actively bleeding, is anticoagulated or on blood thinning medications, or has a bleeding disorder
16. Is a member of a vulnerable population such as prisoners, handicapped or mentally disabled persons, or economically or educationally disadvantaged persons
17. In the opinion of the treating physician, has a contraindication listed in the current NanoKnife System User Manual (section 2.3)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Rate of negative in-field biopsy at 12 months | 12 months
  To determine the NanoKnife System's ablation effectiveness by measuring the negative in-field biopsy rate at 12 months
Incidence of adverse events by type and CTCAE v5.0 severity through 12 months | 12 months
  To determine the NanoKnife System's procedural and post-procedural safety profile by evaluation adverse event incidence, type, and severity through 12 months

SECONDARY OUTCOMES:
Rate of negative in-field biopsy at 12 months as defined by the Delphi consensus criterion | 12 months
  Rate of negative in-field biopsy at 12 months as defined by the Delphi consensus criterion of absence of clinically significant disease (≤ 3 mm of Gleason ≤ 6 disease in any biopsy core is insignificant)
Assessment of urinary function by comparison of pre- and post-operative UCLA Expanded Prostate Cancer Index Composite | 12 months
  Assessment of urinary function by comparison of pre- and post-operative UCLA Expanded Prostate Cancer Index Composite (UCLA-EPIC) Urinary Domain and International Prostate Symptom Scores (IPSS) and IPSS Quality of Life2 (IPSS-QoL) scores.
Assessment of erectile function by comparison of pre- and post-operative IIEF-15 potency scores | 12 months
  Assessment of erectile function by comparison of pre- and post-operative 15-Item International Index of Erectile Function (IIEF-15) potency scores.
Effectiveness of therapy by measurement of prostate-specific antigen (PSA) kinetics | 12 months
  Effectiveness of therapy by measurement of prostate-specific antigen (PSA) kinetics including time to PSA nadir.
Assessment of changes in prostate volume | 12 months
  Assessment of changes in prostate volume by comparison of pre-treatment and 12-month prostate volume measured via mpMRI.
Assessment of ablation effectiveness by evaluation of prostate tissue by mpMRI | 12 months
  Assessment of ablation effectiveness by evaluation of prostate tissue by mpMRI at 3 to 10 days post-treatment and at 12 months post-treatment.
Assessment of need for secondary or adjuvant treatment | 12 months
  Assessment of need for secondary or adjuvant treatment following treatment with the NanoKnife System.
Evaluation of subject reported pre- and post-operative Quality of Life | 12 months
  Evaluation of subject reported pre- and post-operative Quality of Life (QoL) using the 5-dimension scale EuroQol (EQ-5D®).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coleman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Arvin George, MD, Principal Investigator — University of Michigan
Locations (17):
- United States (17):
  - University of California Irvine, Orange, California
  - University of Colorado, Aurora, Colorado
  - University of Florida Health, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University Healthsystem, Evanston, Illinois
  - Duly Health and Care, Lisle, Illinois
  - VA Ann Arbor Health Care, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Northwell Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No